CLINICAL TRIAL: NCT02039297
Title: Patient Centered Cloud-based Electronic System: Ambient Warning and Response Evaluation (ProCCESs AWARE)
Acronym: AWARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brian W. Pickering, M.B., B.Ch., Consultant, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 12-007918
Record Dates: First submitted 2014-01-15; First posted 2014-01-17 (Estimated); Last update posted 2017-10-24 (Actual); Status verified 2017-10

CONDITIONS: Critical Illness; Sepsis; Respiratory Failure; Shock; Coma; Bleeding; Trauma
Keywords: AWARE, Checklist, ICU, Outcome, Adults
MeSH Terms: conditions — Critical Illness; Sepsis; Respiratory Insufficiency; Shock; Coma; Hemorrhage; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- No Intervention: Baseline arm (Other): Pre and post design (same arm)
  Interventions: Other: Patient Centered Cloud-based Electronic System: Ambient Warning and Response Evaluation

INTERVENTIONS:
Other: Patient Centered Cloud-based Electronic System: Ambient Warning and Response Evaluation — Computer aided checklist and rounding tool implemented in the Intensive care unit environment
  Other Names: ProCCESs AWARE

SUMMARY:
In this multicenter project, we will introduce AWARE (electronic interface) Using a cloud-based technology . The goal of this project is to improve compliance with best practice through the use of a new acute care interface with built-in tools for error prevention, practice surveillance and reporting (ProCCESs AWARE - Patient Centered Cloud-based Electronic System: Ambient Warning and Response Evaluation).The goal of this project is to develop and test a novel acute care interface with built-in tools for error prevention, practice surveillance, decision support and reporting (ProCCESs AWARE - Patient Centered Cloud-based Electronic System: Ambient Warning and Response Evaluation). In preliminary studies, these novel informatics supports built on an advanced understanding of cognitive and organizational ergonomics, have significantly decreased the cognitive load of bedside providers and reduced medical errors. Using a cloud-based technology, AWARE will be uniformly available on either mobile or fixed computing devices and applied in a standardized manner in medical and surgical ICUs of five geographically diverse acute care hospitals predominantly serving Medicare and Medicaid patients. The impact of ProCCESs AWARE on processes of care and outcomes in study ICUs; expected to enroll more than 10,000 critically ill patients during the study period.

ELIGIBILITY:
Inclusion Criteria:

For the Primary Objective, all critically ill adult patient admitted to an ICU participating in the study will be eligible.

Exclusion Criteria:

For the Primary Objective, all children younger than 18years of age will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7813 (Actual)
Dates: Start 2013-03; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Adherence to process of care | Participants will be followed for the duration of ICU stay, an expected average of 3 days
  Adherence to best practice for daily intensive care rounds. Appropriate shock resuscitation Appropriate sepsis treatment Appropriate mechanical ventilation Appropriate peptic ulcer, deep vein thrombosis and infectious disease prophylaxis etc.

SECONDARY OUTCOMES:
Patient outcomes | Hospital length of stay - 2 weeks
  We will include, ICU length of stay, Hospital length of stay, ICU free days, standardized mortality ratio in ICU and Hospital, Ventilator free days.

OTHER OUTCOMES:
Cost of patient care in ICU and Hospital | Hospital length of stay - 2 weeks
  Cost of patient care in ICU and Hospital derived from medicare data

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pickering, MBBCh, Principal Investigator — Mayo Clinic; Ognjen Gajic, MD, Principal Investigator — Mayo Clinic; Vitaly Herasevich, MD PhD, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Mayo Clinic, Jacksonville, Florida
  - Lawrence Genral Hospital, Lawrence, Massachusetts
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Montefiore Medical Center, The Bronx, New York
  - OU Medical center, Oklahoma City, Oklahoma

IPD SHARING:
Plan to Share IPD: No